CLINICAL TRIAL: NCT01812993
Title: Reversal of the Neurological Deficit in Acute Stroke With the Signal of Efficacy Trial of Auto BPAP to Limit Damage From Suspected Sleep Apnea (Reverse-STEAL): A Multicenter Randomized Study
Brief Title: Reversal of the Neurological Deficit in Acute Stroke With the Signal of Efficacy Trial of Auto BPAP to Limit Damage From Suspected Sleep Apnea
Acronym: Reverse-STEAL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Dr. Jessica Kepplinger, Instructor, Technische Universität Dresden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RES03_2013
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Ischemic Stroke
Keywords: Ischemic stroke, sleep apnea, non-invasive ventilatory treatment
MeSH Terms: conditions — Ischemic Stroke; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): No ventilatory treatment; standard stroke care
- Active (Experimental): Non-invasive ventilatory treatment with auto-BPAP plus standard stroke care
  Interventions: Device: Non-invasive ventilatory treatment with auto-BPAP

INTERVENTIONS:
Device: Non-invasive ventilatory treatment with auto-BPAP
  Arms: Active

SUMMARY:
Although the negative impact of sleep apnea on the clinical course of acute ischemic stroke (AIS) is well known, data regarding non-invasive ventilation in acute patients are scarce. Several studies showed its tolerability, safety and signals-of-efficacy, yet no controlled randomized sequential phase studies currently exist that aim to establish the efficacy of early non-invasive ventilation in AIS patients. The main hypothesis for this study is that early non-invasive ventilation with automated bilevel positive airway pressure (auto-BPAP) positively affects short-term clinical outcomes in AIS patients. This is a multicenter, prospective, randomized, controlled, third rater-blinded, parallel-group trial. Patients with AIS with proximal arterial obstruction and clinically suspected sleep apnea will be randomized to standard or standard stroke care plus auto-BPAP. Auto-BPAP will be initiated within 24 hours from stroke onset and performed for a maximum of 48 hours during diurnal and nocturnal sleep. Patients will undergo cardiorespiratory polygraphy between day 3 and 5 to assess sleep apnea. The primary endpoint is any early neurological improvement on the NIHSS at 72 hours from randomization. Safety, tolerability, short-term and 3 months functional outcomes are assessed as secondary endpoints by un-blinded and blinded observers respectively. This study will provide data to power a subsequent phase III study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 - 80 years;
* Clinical suspicion of an AIS (measurable or fluctuating neurological deficit with a National Institutes of Health Stroke Scale [NIHSS] ≥ 4 points) within 24 hours from symptom-onset;
* Extracranial (internal carotid artery) or intracranial (internal carotid artery; middle/anterior/posterior cerebral arteries) ≥ 50% stenosis, near-occlusion or occlusion diagnosed by ultrasound, computed tomography angiography (CTA) or magnetic resonance angiography (MRA), corresponding to acute neurological deficit;
* High-risk of having sleep apnea (classified by the Berlin sleep apnea questionnaire); or history of known sleep apnea; or witnessed repetitive apnea episodes during sleep or somnolence during hospitalization;
* Written informed consent by participants; alternatively by proxy or two physicians when not obtainable by patient or proxy (according to local regulations).

Exclusion Criteria:

* Perceived course towards the malignant middle cerebral artery infarction;
* Immediate or perceived need for intubation;
* Known sleep apnea currently on non-invasive ventilatory treatment;
* Standard contraindications for non-invasive ventilatory treatment;
* Pre-morbid modified Rankin scale (mRS) score ≥ 3;
* Severe comorbidities (i.e., severe heart failure, severe obstructive lung disease, active malignant disease, severe dementia);
* Pregnant and breast feeding women;
* Participation in another clinical trial other than standard-of-care registry.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Early neurological recovery | 72+12 hours from randomization
  Early neurological recovery will be assessed as any improvement on the NIHSS score at 72+12 hours from randomization

SECONDARY OUTCOMES:
Tolerability | During treatment with auto-BPAP; up to 48 hours
  Tolerability will be assessed by patients' adherence to auto-BPAP (defined as tolerating the treatment during sleep or somnolence for at least 4 hours continuously)
Safety | During treatment with auto-BPAP; up to 72 hours from randomization
  Safety will be assessed by:
  (i) frequency of serious adverse events (i.e., aspiration, aspiration pneumonia defined as combined radiologic, white blood count and clinical findings, respiratory failure with/without intubation) during treatment period that in the opinion of the study physician are causatively and timely (for a maximum of 72 hours from treatment initiation) related to auto-BPAP and all deaths during hospital stay. For comparison, patients in the control group will be monitored for respiratory complications within 72 hours from randomization; (ii) frequency of all complaints and possible side effects of auto-BPAP (i.e., local irritation of skin/mucosa, mucosal dryness, nausea/vomiting); (iii) any concerns by hospital nursing staff will be documented as adverse events since patients will be under standard of care repeated assessments set by admission protocols and treating physicians.
Signal-of-efficacy | 24 hours; discharge; 90 days from randomization
  Signal-of-efficacy:
  Clinical and functional outcomes will be assessed by:
  (i) frequency of neurological deterioration (increase in baseline NIHSS score ≥4 points) at 24, 48 and after 72 hours from randomization by blinded observers; (ii) frequency of early neurological improvement (decrease in baseline NIHSS score ≥4 points) at 24, 48 and after 72 hours from randomization by blinded observers; (iii) good functional outcome (mRS score 0-2) at discharge and at 3 months by blinded observers; (iv) any TIA or new ischemic stroke during hospitalization or within 3 months of protocol initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei V. Alexandrov, MD, Principal Investigator — University of Alabama at Birmingham; Ulf Bodechtel, MD, Principal Investigator — University of Technology Dresden; Jessica Kepplinger, MD, Principal Investigator — University of Technology Dresden
Locations (4):
- University of Tennessee Health Science Center, Department of Neurology, Memphis, Tennessee, United States
- Department of Neurology, General Hospital Linz (AKH), Linz, Austria
- International Clinical Research Center, St. Anne's University Hospital Brno, Brno, Czechia
- Dresden University Stroke Center, University of Technology Dresden,, Dresden, Germany

REFERENCES:
- [Derived] Barlinn K, Jakubicek S, Siepmann T, Chernyshev OY, Pallesen LP, Wienecke M, Hermann W, Graehlert X, Alexandrov AW, Vosko M, Puetz V, Reichmann H, Bodechtel U, Mikulik R, Barlinn J, Alexandrov AV. Autotitrating Bilevel Positive Airway Pressure in Large Vessel Steno-Occlusive Stroke Patients With Suspected Sleep Apnea: A Multicenter Randomized Controlled Study. Front Neurol. 2021 Apr 13;12:667494. doi: 10.3389/fneur.2021.667494. eCollection 2021. PMID 33927689
- [Derived] Kepplinger J, Barlinn K, Kolieskova S, Shahripour RB, Pallesen LP, Schrempf W, Graehlert X, Schwanebeck U, Sisson A, Zerna C, Puetz V, Reichmann H, Albright KC, Alexandrov AW, Vosko M, Mikulik R, Bodechtel U, Alexandrov AV. Reversal of the neurological deficit in acute stroke with the signal of efficacy trial of auto-BPAP to limit damage from suspected sleep apnea (Reverse-STEAL): study protocol for a randomized controlled trial. Trials. 2013 Aug 13;14:252. doi: 10.1186/1745-6215-14-252. PMID 23941576